CLINICAL TRIAL: NCT06549036
Title: Randomized Trial of Veteran Peer Navigators to Promote Shared Decision Making for PSA Screening
Brief Title: Veteran Peer Navigators to Promote Shared Decision Making for PSA Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IIR 22-090; I01HX003622-01A2 (NIH)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Prostate-Specific Antigen; shared decision making
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Veterans randomized to the intervention arm will receive a decision aid in the mail along with decision coaching on PSA screening from a Veteran Veteran-peer-navigator decision coach. The intervention will be administered prior to the Veteran patient's appointment with the provider.
  Interventions: Behavioral: Veteran Peer Decision Coaching Session for PSA Screening
- Control Group (No Intervention): Veteran patients in the control arm will receive a decision aid alone in the mail without any additional counseling prior to their office visit.

INTERVENTIONS:
Behavioral: Veteran Peer Decision Coaching Session for PSA Screening — Veterans in the intervention arm will review the content of the mailed DA, including the values clarification exercise, with the Veteran PDC. Veteran PDC Counseling includes: 1) a structured interview with the patient that focuses on determining his understanding of his prostate cancer risk, his screening options, and his goals and values related to his decision making and 2) role playing exercises to improve SDM skills.
  Other Names: PDC Intervention
  Arms: Intervention Group

SUMMARY:
The project will investigate the efficacy of a Veteran-peer-navigator-led decision coaching (PDC) program to promote Shared Decision Making (SDM) for prostate cancer screening among Veterans at the Veterans Health Administration (VA). Prostate cancer is commonly screen detected using PSA, a non-specific test which has led to modest population-level survival benefits at the cost of over-detection of low-risk disease. This trade off in outcomes is ideally addressed using SDM which can be challenging to implement in time constrained primary care office visits. The investigators propose the evaluation of a PDC intervention to promote SDM for PSA screening to improve both access and quality of care for Veterans. The investigators results will enhance understanding of the efficacy, cost-effectiveness, and sustainability of PDC interventions for SDM promotion across communication formats in the VA. Lessons learned through this proposal will not only improve quality of care for PSA screening but also will suggest a paradigm for dissemination of SDM across preventive services.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-cutaneous malignancy among men in the United States, accounting for one third of new cancer diagnoses in VA. Prostate Cancer is commonly detected using prostate-specific antigen (PSA), a non-specific test whose use in prostate cancer screening has led to modest population-level survival benefits at the cost of over-detection of low-risk disease. Recognizing this trade off, USPSTF and VHA Clinical Preventive Services recommend a Shared Decision Making (SDM) approach to PSA screening. Regardless of whether they ultimately elect PSA screening or not, patients should discuss the best evidence for and against it with clinicians and be supported to make high quality decisions. In spite of broad support for these recommendations, SDM is challenging to implement because primary care providers see it as too time consuming and have insufficient training and support to perform it. Moreover, primary care office visits are notoriously too brief to address the multitude of recommended, beneficial preventive interventions. There is an urgent need to incorporate SDM paradigms into routine VA clinical practice. An ideal intervention accomplishing this would improve decision quality at low cost and be acceptable to Veterans and clinicians.

The primary challenge to implementing routine PSA SDM counseling is clinic workflow. One solution may be to enlist non-clinician healthcare team members to offer SDM counseling. Decision coaches can provide non-directive support to help patients weigh options, prepare for provider discussions, and implement decisions. Decision coaches improve knowledge and promote SDM. In a pilot program, the investigators group trained lay health workers as decision coaches to counsel Black men considering PSA screening in a non-VA community care setting. There is an urgent need to expand this approach to all men considering PSA screening and adapt it to the VA setting. The investigators propose training Veteran peers, who are well-known to promote healthful behaviors among Veterans, to be decision coaches to promote SDM among Veterans considering PSA screening. This peer-led approach may provide excellent counseling at acceptable cost and decreased clinician burden.

The objective of this study is to test the efficacy of a Veteran-peer-navigator-led decision-coaching program (PDC) to facilitate SDM for PSA screening at VA NY Harbor. The investigators will randomize Veterans seeking primary care to receive 1) a standard of care screening decision aid (DA) along with PDC on PSA screening (intervention), or 2) the same DA without counseling (control). The outcomes of interest are decision quality, PSA utilization, acceptability and cost of the PDC program with the goal of future system-wide dissemination. Additionally, since VA is dedicated to promoting health equity through telehealth, the investigators will explore the effects of patient race (Black versus non-Black) and communication format (in-person versus telehealth).

ELIGIBILITY:
Inclusion Criteria:

Veteran patient participants:

* Age 40-69 years old
* Veteran
* Male
* Attending VANYHHS-Manhattan for routine primary care appointment

Providers:

* Primary care provider at VA New York Harbor Healthcare System (VANYHHS)
* Caring for patients that fit inclusion criteria

Exclusion Criteria:

Veteran Patients:

* Patients seen within 9 months of other PSA tests
* Patients seen within 180 days after primary diagnosis of urinary obstruction, prostatitis, hematuria, other disorder of prostate, unexplained weight loss, or lumbar back pain
* Patients with a prior diagnosis of prostate cancer (ICD-10-CM C61)
* Patients visiting their provider for any indication other than a well-visit appointment

Providers:

- Providers who do not treat adult male patients (e.g. OB/Gyns, pediatricians)

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be male based on inclusion criteria. Providers do not have any gender eligibility requirements.
Enrollment: 228 (Estimated)
Dates: Start 2026-03-23 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict | Up to 3 months
  The 16-item Decisional Conflict Scale (DCS) measures Veterans' perceptions of 1) uncertainty in choosing options, 2) feelings of having adequate knowledge and clear values, and 3) effective decision making. DCS is scored on a 5-point Likert scales with scores ranging from 0 (no decisional conflict) to 100 (extremely high decisional conflict)
Patient Knowledge Survey Score | Day 1
  The Patient Knowledge Survey comprises of 12-items assessing prostate cancer and PSA screening knowledge. Respondents provide an answer of "True", "Unsure", or "False". The total score is the sum of correct responses and ranges from 0 - 12 with higher scores indicating greater knowledge levels.
Decision Quality Score | Day 1
  Decision quality will be measured through 3 domains: 1) decisional conflict 2) being informed (e.g. accurate understanding about screening and its risks and benefits) and 3) making preference-concordant decisions (i.e. treatment consistent with patient preferences). The Decision Quality Balance Scale consists of 12 questions (6 Pros and 6 Cons of testing) scored on a 5 point Likert scale (Strongly Disagree to Strongly Agree) that represents the relative strengths of the pros versus the cons and ranges from -24 to +24. A high quality decision is when patients are both well-informed and making preference-concordant decisions (i.e. treatment consistent with patient preferences as determined by responses to survey questions).
Prostate-specific Antigen (PSA) Screening Rates | Up to Month 3
  Percentage of participants who receive at least one PSA screening test. Screening data is collected through patient self-report and electronic health record data.
Percentage of Participants Who Make Informed Choice (Knowledge Survey + Measure of Informed Choice Attitudes Scale) | Day 1
  The percentage of participants who make an informed choice to either undergo or decline PSA testing. Informed choices are those in which:
  1. Men with good knowledge and positive measure of informed choice attitudes (> or = 22) choose to undergo the test OR 2) Men with good knowledge but negative measure of informed choice attitudes (<22) towards the test, do not undergo the test.
Measure of Informed Choice Attitudes Scale | Day 1
  The measure of Informed Choice evaluates the screening decision. The 4-item measure consists of items assessing knowledge, attitude towards the screening test, and a record of test uptake. The questions are graded on a 7 point Likert-type scale (1 to 7) with scores ranging from 4 to 28. The median of 22 was taken to classify men's attitudes as positive or negative, with scores 22 or above indicating positive attitudes, and those below 22 indicating negative attitudes.

SECONDARY OUTCOMES:
Combined Outcome Measure for Risk communication And treatment Decision making Effectiveness (COMRADE) | Day 1
  Combined Outcome Measure for Risk communication And treatment Decision making Effectiveness (COMRADE) is a 20-item measure validated for clinical encounters with sub-scales in 1) satisfaction with physician communication and 2) patient confidence in the decision. The scale is graded on a 5 point Likert scale (1 to 5) with a range from 1 to 100 maximum. Higher scores indicate higher satisfaction with communication.
Doctor-Patient Communication Survey | Day 1
  The Questionnaire Concerning Doctor-Patient Communication Skills is a validated 19 item scale that captures process (greeting, listening) and content (explanations and next steps) aspects of the visit from the provider's and patient's perspectives. The questions are scored on a 5-point Likert scale (1 Strongly Disagree to 5 Strongly Agree) with Higher scores (4-5) indicating satisfaction with provider communication
Decision Self-Efficacy | Day 1
  The Decision Self-Efficacy Scale is an 11 item scale measuring self-efficacy to perform informed decision making (e.g. getting needed information, asking questions, expressing opinions, and asking for advice). The questions are scored on a 5-point Likert scale (0 Strongly Disagree to 4 Strongly Agree) and range from 0 (not at all confident) to 100 (very confident).
Self-efficacy for Communicating with Provider | Day 1
  Perceived Efficacy in Patient-Physician Interactions is a 10-item scale measuring self-efficacy for communicating with a provider. The questions are scored on a 5-point Likert scale (1 Not at all confident to 5 Very confident) with a range of possible scores from 10 to 50 (highest patient perceived self-efficacy for communicating with provider).
Satisfaction with Decision Scale | Up to 3 Months
  The SWD is a 6-item measure assessing patient satisfaction with their decision and the decision making process. The questions are scored on a 5-point Likert scale (1 Strongly Disagree to 5 Strongly Agree). Higher scores indicate higher satisfaction with decision (scores range from 1-5).
Decisional Regret Scale | Up to 3 Months
  The Decisional Regret Scale is a validated, 5-item scale measuring regret or remorse following a health care decision. Questions are scored on a 5-point Likert scale (5 Strongly Disagree to 1 Strongly Agree). Scores range from 0 (means no regret) to 100 (means high regret).

CONTACTS AND LOCATIONS:
Overall Officials: Danil V Makarov, MD MHS, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright Nunes J, Kerr E, Ojo A, Powell C, Fan A, Brinley FJ, Devine A, Ellies T, Grzyb K, Garcia-Guzman L, Nakai T, Oliverio A, Chen E, Fagerlin A. Patient Education for CKD and Decision Support in Primary Care: Findings From the EPIK Pilot Study. Am J Kidney Dis. 2025 Mar;85(3):284-292. doi: 10.1053/j.ajkd.2024.10.005. Epub 2024 Dec 14. PMID 39675547